CLINICAL TRIAL: NCT05452213
Title: CAPTOR-BC: Comprehensive Analysis of Spatial, Temporal and Molecular Patterns of Ribociclib Efficacy and Resistance in Advanced Breast Cancer Patients
Brief Title: Comprehensive Analysis of Spatial, Temporal and Molecular Patterns of Ribociclib Efficacy and Resistance in Advanced Breast Cancer Patients
Acronym: CAPTOR-BC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institut fuer Frauengesundheit (Other)
Collaborators: AGO Breast Study Group e.V. (Unknown); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFG-01-2022
Record Dates: First submitted 2022-06-28; First posted 2022-07-11 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Neoplasm Female; Breast Cancer Female; HER2-negative Breast Cancer; Hormone Receptor-positive Breast Cancer; Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Intervention Model Description: One-arm, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ribociclib (Experimental)
  Interventions: Drug: Ribociclib

INTERVENTIONS:
Drug: Ribociclib — All patients will receive ribociclib in combination with standard endocrine therapy according to the current SmPC and local in-house standard.
  Ribociclib will be administered once daily for 21 consecutive days followed by 7 days off treatment (28-day cycle). The daily dose is 600 mg/day.
  Ribociclib and standard of care endocrine treatment will be prescribed and administered according to investigator's discretion.

SUMMARY:
This is a single-arm, open-label phase IV study of patients with advanced HR+/HER2- breast cancer who are treated first line with ribociclib and standard of care endocrine treatment according to SmPC.

DETAILED DESCRIPTION:
This is a prospective, multicenter, phase IV, one-arm, open-label clinical trial investigating patients treated with ribociclib and standard of care endocrine therapy for hormone receptor positive (HR+) / human epidermal growth factor receptor negative (HER2-) advanced breast cancer in the first therapy line. Patients eligible for this trial will receive on-label ribociclib according to Summary of Product Characteristics (SmPC) and as well as the specified inclusion/exclusion criteria.

The survival rates for progression-free survival (PFS) and overall survival (OS) at month 12 are the co-primary objectives. Quality of life and toxicity are secondary objectives. Additionally, there is a comprehensive biomarker discovery and validation program included into the study.

A total of 1000 patients are planned to be enrolled into this trial in 75 trial sites in Germany.

Biomarkers will be evaluated before, during and after treatment or at progression. A comprehensive biospecimens sampling will be done to enable translational research projects and evaluation of potential biomarkers within circulation tumor desoxyribonucleic acid (ctDNA), circulating tumor ribonucleic acid (ctRNA), formaldehyde-fixed paraffin-embedded tissue (FFPE) tissue, Serum, Plasma and circulating immune cells

ELIGIBILITY:
Inclusion Criteria:

1. Indication for treatment with ribociclib in combination with endocrine therapy in the locally advanced or 1st line metastatic therapy setting according to SmPC. (Previous treatment with cycline dependent kinase 4/6 (CDK4/6) inhibitors is allowed in the adjuvant setting)
2. Written informed consent prior to beginning of trial specific procedures
3. Subject must be female and aged ≥ 18 years on the day of signing informed consent
4. Locally advanced or metastatic breast cancer not amenable to curative treatment
5. Patient has HER2-negative breast cancer confirmed by local laboratory defined as a negative in situ hybridization test or an immunohistochemistry (IHC) status of 0 or 1+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required to confirm the HER2-negative status (based on the most recently analyzed tissue sample tested by a local laboratory
6. Histologically confirmed estrogen receptor (ER) positive and/ or progesterone receptor (PgR) positive breast cancer determined by core biopsy according to local in-house standard.
7. corrected QT (QTcF) interval < 450 ms
8. Adequate organ function amenable for treatment with ribociclib as assessed by local laboratory
9. Women of childbearing potential must have a negative urine or serum pregnancy test within 72 h prior to study entry and be willing to use highly effective method of contraception for course of the trial through 21 days after the last dose of trial treatment.
10. Patient must be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Concurrent participation in a study with an investigational agent/device or within 14 days of study entry or 5 half-lives of the respective investigational agent/device, whichever is longer
2. Patients who are not treated for advanced HR+, HER2- breast cancer in the first line therapy setting.
3. Patient not eligible for treatment with ribociclib according to SmPC or investigator's discretion
4. Patients who are pregnant or lactating.
5. Patients with existing or patients who are at significant risk of developing corrected QT interval (QTc) prolongation. This includes

   * patients with long QT syndrome
   * uncontrolled or significant cardiac disease, including recent myocardial infarction, congestive heart failure, unstable angina and bradyarrhythmia
   * electrolyte abnormalities
6. Patients with known hypersensitivity to the active substance of ribociclib, soya, peanut or any other of the excipients of ribociclib.
7. Patients with active systemic infections (for example, bacterial infection requiring intravenous antibiotics at time of initiating study treatment, fungal infection, or detectable viral infection requiring systemic therapy) or viral load (such as known human immunodeficiency virus positivity or with known active hepatitis B or C, for example, hepatitis B surface antigen positive).
8. Patients with serious preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (such as severe renal impairment, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in clinically significant diarrhea).
9. Patient who do not agree to collection of biospecimens samples (blood, stool, tissue)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
12-month PFS rate | 12 months
  The rate for progression-free survival at month 12 will be calculated.
12-month OS rate | 12 months
  The rate for overall survival at month 12 will be calculated.

SECONDARY OUTCOMES:
24-month PFS rate | 24 months
  The rate for progression-free survival at month 24 will be calculated.
24-month OS rate | 24 months
  The rate for overall survival at month 24 will be calculated.
36-month PFS rate | 36 months
  The rate for progression-free survival at month 36 will be calculated.
36-month OS rate | 36 months
  The rate for overall survival at month 36 will be calculated.
Median progression-free survival | From date of enrollment until first documented progression or date of death from any cause or regular end of study (up to 24 months) whichever is first.
  Median progression-free survival will be estimated if achieved at the end of study
Median overall survival | From date of enrollment until date of death from any cause or regular end of study (up to 24 months) whichever is first.
  Median overall survival will be estimated if achieved at the end of study
Health related quality of life (FACT-G) | Collected before start of trial treatment, at 3 months and every 6 months afterwards until end of study up to 24 months
  Health related quality of life as assessed by FACT-G questionnaire (Functional Assessment of Cancer Therapy - General) Min 0, Max 108, The higher the score, the better the QoL.
Health related quality of life (FACT-B) | Collected before start of trial treatment, at 3 months and every 6 months afterwards until end of study up to 24 months
  Health related quality of life as assessed by FACT-B questionnaire (Functional Assessment of Cancer Therapy - Breast Cancer) Min 0, Max 148, The higher the score, the better the QoL.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | All adverse events will be recorded from signing informed consent through 30 days following cessation of treatment or until the last study visit
  The safety endpoints for the study will include rate of adverse events (AE), serious adverse events (SAEs) and fatal SAEs, causality and outcome of AE/SAEs, rate of treatment discontinuations and reasons, Changes in vital signs, laboratory values etc. Grading of AE/SAEs will be based on NCI CTCAE v5.0.

OTHER OUTCOMES:
Correlation of genome wide genetic biomarkers with progression-free survival | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Genome wide genetic biomarkers will be assessed by whole genome sequencing and/ or panel sequencing from blood samples.
Correlation of genome wide genetic biomarkers with overall survival | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Genome wide genetic biomarkers will be assessed by whole genome sequencing and/ or panel sequencing from blood samples.
Correlation of genome wide genetic biomarkers with quality of life | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Genome wide genetic biomarkers will be assessed by whole genome sequencing and/ or panel sequencing from blood samples.
Correlation of genome wide genetic biomarkers with ribociclib side effects | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Genome wide genetic biomarkers will be assessed by whole genome sequencing and/ or panel sequencing from blood samples.
Correlation of genome wide gene expression biomarkers with progression-free survival | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Genome wide genetic biomarkers will be assessed by whole genome sequencing and/ or panel sequencing from blood samples.
Correlation of genome wide gene expression biomarkers with overall survival | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Genome wide genetic biomarkers will be assessed by whole genome sequencing and/ or panel sequencing from blood samples.
Correlation of genome wide gene expression biomarkers with quality of life | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Genome wide genetic biomarkers will be assessed by whole genome sequencing and/ or panel sequencing from blood samples.
Correlation of genome wide gene expression biomarkers with ribociclib side effects | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Genome wide genetic biomarkers will be assessed by whole genome sequencing and/ or panel sequencing from blood samples.
Correlation of genome wide tumor mutational patterns assessed from formalin-fixed paraffin embedded tumor material with progression-free survival | Measured from biomaterial collected at baseline and at the time of tumor progression
  Tumor DNA will be either isolated from FFPE tissue (primary tumor or metastasis) or from Plasma samples (STRECK cfDNA Tube). DNA will be analyzed by whole genome sequencing and/or panel sequencing.
Correlation of genome wide tumor mutational patterns assessed from formalin-fixed paraffin embedded tumor material with overall survival | Measured from biomaterial collected at baseline and at the time of tumor progression
  Tumor DNA will be either isolated from FFPE tissue (primary tumor or metastasis) or from Plasma samples (STRECK cfDNA Tube). DNA will be analyzed by whole genome sequencing and/or panel sequencing.
Correlation of genome wide tumor mutational patterns assessed from formalin-fixed paraffin embedded tumor material with quality of life | Measured from biomaterial collected at baseline and at the time of tumor progression
  Tumor DNA will be either isolated from FFPE tissue (primary tumor or metastasis) or from Plasma samples (STRECK cfDNA Tube). DNA will be analyzed by whole genome sequencing and/or panel sequencing.
Correlation of genome wide tumor mutational patterns assessed from formalin-fixed paraffin embedded tumor material with ribociclib side effects | Measured from biomaterial collected at baseline and at the time of tumor progression
  Tumor DNA will be either isolated from FFPE tissue (primary tumor or metastasis) or from Plasma samples (STRECK cfDNA Tube). DNA will be analyzed by whole genome sequencing and/or panel sequencing.
Correlation of genome wide tumor mutational patterns assessed from ctDNA biomarkers with progression-free survival | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Germline DNA will be isolated from one EDTA blood samples obtained within the study. DNA will be analyzed by whole genome sequencing and/or panel sequencing.
Correlation of genome wide tumor mutational patterns assessed from ctDNA biomarkers with overall survival | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Germline DNA will be isolated from one EDTA blood samples obtained within the study. DNA will be analyzed by whole genome sequencing and/or panel sequencing.
Correlation of genome wide tumor mutational patterns assessed from ctDNA biomarkers with quality of life | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Germline DNA will be isolated from one EDTA blood samples obtained within the study. DNA will be analyzed by whole genome sequencing and/or panel sequencing.
Correlation of genome wide tumor mutational patterns assessed from ctDNA biomarkers with ribociclib side effects | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Germline DNA will be isolated from one EDTA blood samples obtained within the study. DNA will be analyzed by whole genome sequencing and/or panel sequencing.
Correlation of changes in the genome wide tumor mutational patterns assessed from ctDNA biomarkers with progression-free survival | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Germline DNA will be isolated from one EDTA blood samples obtained within the study. DNA will be analyzed by whole genome sequencing and/or panel sequencing.
Correlation of changes in the genome wide tumor mutational patterns assessed from ctDNA biomarkers with overall survival | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Germline DNA will be isolated from one EDTA blood samples obtained within the study. DNA will be analyzed by whole genome sequencing and/or panel sequencing.
Correlation of changes in the genome wide tumor mutational patterns assessed from ctDNA biomarkers with quality of life | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Germline DNA will be isolated from one EDTA blood samples obtained within the study. DNA will be analyzed by whole genome sequencing and/or panel sequencing.
Correlation of changes in the genome wide tumor mutational patterns assessed from ctDNA biomarkers with ribociclib side effects | Measured from biomaterial collected at baseline, 2 weeks, 3 months, 6 months, 12 months, 18 months or at the end of treatment in case treatment is stopped irregularly.
  Germline DNA will be isolated from one EDTA blood samples obtained within the study. DNA will be analyzed by whole genome sequencing and/or panel sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Fasching, MD, Prof., Study Chair — Department of Gynecology and Obstetrics, Erlangen University Hospital; Tanja Fehm, MD, Prof., Study Chair — Department of Gynecology/Obstetrics |University Hospital Düsseldorf, Germany; Andreas Schneeweiss, MD, Prof., Study Chair — National Center for Tumor Diseases (NCT) | Heidelberg University Hospital and German Cancer Research Center
Locations (52):
- Germany (52):
  - Department of Gynecology and Obstetrics, Erlangen University Hospital, Erlangen, Bavaria
  - Department of Gynecology and Obstetrics, University Medicine Mainz, Mainz, Hesse
  - Department for Gynecology and Obstetrics, Marienhospital Bottrop gGmbH, Bottrop, North Rhine-Westphalia
  - Klinikum St Marien Amberg, Amberg
  - Onkologie Aschaffenburg, Hämato-Onkologische Schwerpunktpraxis am Klinikum Aschaffenburg, Aschaffenburg
  - Klinik für Hämatologie und Onkologie, Uniklinik Augsburg, Augsburg
  - University Hospital Augsburg, Augsburg
  - Frauenklinik des Klinikums Bamberg, Bamberg
  - MediOnko GbR, Berlin
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Zentrum für ambulante Hämatologie und Onkologie (ZAHO) an der Robert-Janker-Klinik, Bonn
  - Klinik für Gynäkologie, Gynäkoonkologie und Senologie Klinikum Bremen-Mitte, Bremen
  - Klinikum Chemnitz gGmbH, Klinik für Frauenheilkunde und Geburtshilfe, Chemnitz
  - Kliniken Der Stadt Köln gGmbH, Cologne
  - Carl-Thiem-Klinikum Cottbus, Cottbus
  - Staedtisches Klinikum Dessau, Gynecology and Obstetrics, Dessau
  - Universitäts-Frauenklinik Carl Gustav Carus Universität Dresden, Dresden
  - Universitaetsklinikum Duesseldorf AöR, Düsseldorf
  - Universitaetsklinikum Essen AöR, Gynecology and Obstetrics, Essen
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Agaplesion Frankfurter Diakonie Kliniken gGmbH, Gynecology and Obstetrics, Frankfurt am Main
  - Universitäts-Frauenklinik Frankfurt, Frankfurt am Main
  - Universitäts-Frauenklinik Freiburg, Freiburg im Breisgau
  - Medizinisches Versorgungszentrum Onkologie Georgsmarienhütte und Bramsche, Georgsmarienhütte
  - Universitäts-Frauenklinik Hamburg-Eppendorf, Hamburg
  - Mammazentrum Hamburg am Krankenhaus Jerusalem, Hamburg
  - Nationales Centrum für Tumorerkrankungen, Universitätsklinikum Heidelberg Abteilung für Gynäkologie und Geburtshilfe, Heidelberg
  - Frauenklinik, SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Staedtisches Klinikum Karlsruhe gGmbH, Gynecology and Obstetrics, Karlsruhe
  - University Medical Centre Schleswig-Holstein, Gynecology and Obstetrics, Kiel
  - ZAGO-Zentrum für ambulante gynäkologische Onkologie, Krefeld
  - Klinikum Kulmbach, Kulmbach
  - VK&K Studienzentrum Landshut am Lakumed Klinikum Landshut-Achdorf, Landshut
  - Praxis Dr. Müller MVM GmbH, Studienzentrum UnterEms, Leer
  - Universitäts-Frauenklinik Leipzig, Leipzig
  - Ev. Krankenhaus Bethesda Mönchengladbach, Mönchengladbach
  - Hämatologie Onkologie Gemeinschaftspraxis Pasing, Munich
  - MVZ Nordhausen gGmbH, Nordhausen
  - Klinikum Nürnberg, Nuremberg
  - Frauenklinik, Medius Klinik Nürtingen, Nürtingen
  - Gemeinschaftspraxis für Hämatologie und Onkologie GbR, Ravensburg
  - Frauenklinik, Diakoniekrankenhaus Rotenburg, Rotenburg (Wümme)
  - Leopoldina Krankenhaus der Stadt Schweinfurt gGmbH, Schweinfurt
  - Schwerpunktpraxis für Hämatologie, Onkologie und Magen-Darm Diagnostik, Singen
  - Onkologische Schwerpunktpraxis Speyer, Speyer
  - Klinikum Stuttgart, Stuttgart
  - Onkologie Rheinsieg, Praxisnetzwerk Hämatologie und internistische Onkologie, Troisdorf
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitäts-Frauenklinik Ulm, Ulm
  - MVZ Nordoberpfalz, Weiden
  - Medizinische Studiengesellschaft Nord-West GmbH, Westerstede
  - Rems-Murr Kliniken Winnenden, Winnenden

IPD SHARING:
Plan to Share IPD: No